CLINICAL TRIAL: NCT07292467
Title: Evaluation of the Benefits of Shampoo During 4 Weeks of Treatment and After 24 Weeks With 1 Application Per Week (Maintenance Phase) on Subjects With Moderate to Severe Dandruff and Severe Itching State.
Brief Title: Evaluation of the Benefits of Shampoo During 4 Weeks of Treatment and After 24 Weeks
Status: Active, not recruiting | Type: Observational
Sponsor: Vichy Laboratoires (Industry)
Responsible Party: Sponsor
Other Study IDs: VCY 25-001
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Dandruff
MeSH Terms: conditions — Dandruff | interventions — selenium disulfide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Shampoo
  Interventions: Other: Selenium disulfide

INTERVENTIONS:
Other: Selenium disulfide — 1% SeS2

SUMMARY:
The goal of this study to evaluate the efficacy of shampoo after 4 weeks (treatment phase) and after 5 weeks, 8 weeks, 10 weeks, 12 weeks, 16 weeks, 20 weeks and 24 weeks with 1 application per week (maintenance phase) on subjects with moderate to severe dandruff and severe itching state.

Participants will:

Apply investigationnal products 3 time a week during 4 weeks and investigational product once a week and neutral product twice a week during 24 weeks Visit the center 10 times during the study for evaluations Keep a diary of their discomfort and the number of times they use the investigational products

DETAILED DESCRIPTION:
=> after 4 weeks (treatment phase) and 5 weeks, 8 weeks, 10 weeks, 12 weeks, 16 weeks, 20 weeks and 24 weeks with 1 application per week (maintenance phase)

Primary objective :

• To evaluate the reduction of total dandruff ( adherent and non-adherent)

Secondary objectives:

* To evaluate the Quality of Life (QoL) evolution
* To evaluate the reduction of discomfort (itching, stinging, burning sensation)
* To evaluate the reduction of scales
* To assess the cosmetic properties of investigational product
* To assess the tolerance of investigational product

ELIGIBILITY:
Inclusion Criteria:

* At baseline: A moderate to severe level of squames: Total squames score (adherent + non-adherent) ≥ 4 (ranging from 0 to 10) including an adherent squames score ≥ 2.5 (ranging from 0 to 5) and no limit for non-adherent squames score at inclusion (The groups must be balanced to ensure an equitable distribution)
* All types of scalp.
* Any phototype
* Questionnaire inclusion: Food habits and sleep (at least 30 vols per item, a subject can be included in both groups)
* Severe itching score ≥ 7
* Subject with hair length > 2 cm.
* Subject having received the information about the study modalities and having given his/her written consent and having signed the "informed consent form" specific for this study, in accordance with the corresponding procedure.
* Subject usually using a shampoo 3 times a week and accepting to follow a rate of 3 times a week during the whole study period.
* Subject agreeing not to use any other hair product other than the ones provided for the study (till the end of study); in particular:

  * no styling product (tonic, spray, lotion, foam) three days before the study visit.
  * no treating haircare product (conditioner, hair mask, non-rinsed hair care product, oil….).
  * no anti-scales products (whatever the type: shampoo, treatment...).
  * no hair coloring or hair bleaching within one week prior to any study visit.
* Subject agreeing not to have a short haircut during the entire study period.
* Subjects in good general and mental health in the opinion of the investigator
* Subjects demonstrating understanding of the study procedures, restrictions, and willingness to participate as evidenced by voluntary written informed consent and having received a signed and dated copy of the informed consent form
* Subjects who have agreed to comply with the procedures and requirements of the study and to attend the scheduled assessment visits

Exclusion Criteria:

* Subject with scalp psoriasis
* Subject with more than 60% of white hair influencing the scoring of scales.
* Subject who has skin marks on the scalp that could interfere with the assessment (pigmentation trouble, scar elements…).
* Subject with alopecia in vertex (stage > IIIa Hamilton and > I Ludwig)
* Subject who has used topic treatment for the scalp (anti-hair loss, soothing…) during the last three weeks before the start of the study.
* Subject who has used products for the scalp (dyeing, bleaching, permanent waving and straightening …) within the three weeks prior to the study.
* Subject with history of allergy and/or reactions to latex.
* Subject who has taken:

  * Corticoids (local or per os) within 2 weeks before the study entry
  * Anti-histaminic, anti-fungal, non-steroidal anti-inflammatory, immunosuppressive orlithium-based drugs less than 1 month before the study entry,
  * retinoid acid (local or per os) since less than 6 months before study entry.
* Subject practicing regularly water sport and/or having regular sauna sessions.
* Subject exposed to the sun or UV rays in an excessive way during the last month (according to the investigator).
* Pregnancy, breastfeeding, childbearing potential without adequate contraception, or irregular menstrual cycles.
* History of drug or alcohol abuse
* History or suspicion of unreliability, poor cooperation or noncompliance with medical treatment
* Topical treatment of the scalp with other antifungal medication or with corticosteroids in the last 3 weeks before the start of the study.
* Systemic use of erythromycin, tetracycline or any of its derivatives, trimethoprim/sulfamethoxazole, or metronidazole within 28 days before the start of the study
* Subject with personal history of allergy and/or adverse reactions to cosmetic products containing surfactant agents (soaps, shower gel, conditioner …)
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol
* Clinical signs and/or history of immunosuppression
* Severe disease (e.g. cancer, cardiac infarct, unstable angina pectoris pectoris)
* Treatment with any other investigational drug in the 4 weeks prior to study entry
* Employee of the sponsor or the study site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe dandruff and severe itching state in Phoenix in Mauritius
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Dandruff evaluation (non adherent and adherent) | Day 0, Week 4, Week 9, Week 12, Week 14, Week 16, Week 20, Week 24 and Week 28
  Total score of dandruff = score of adherent and non adherent dandruff, which are 2 scales from 0 to 5 "0 is equivalent to no dandruff and 5 indicates a very large quantity of dandruff.

SECONDARY OUTCOMES:
Self-evaluation by subject of discomfort sensation (stinging, itching, burning sensation) on structured scale; | Day 0, Week 4, Week 9, Week 12, Week 14, Week 16, Week 20, Week 24 and Week 28
  Structured scale 0 to 9 (0 is equivalent to none, positive result and 9 indicates hugely, negative result)
Self-evaluation by subject of dandruff state and greasy aspect on structured scale | Structured scale 0 to 9 (0 is equivalent to none, positive result and 9 indicates hugely, negative result)
  Structured scale 0 to 9 (0 is equivalent to none, positive result and 9 indicates hugely, negative result)
Quality of life questionnaire - Scalpdex | Day 0, Week 4, Week 9, Week 12, Week 14, Week 16, Week 20, Week 24 and Week 28
  Publish questionnaire of quality of life, each item is evaluate with a 5-point scale from 0 (never, positive result) to 100 (always, negative result)
Standardized pictures of the scalp | Day 0, Week 4, Week 9, Week 12, Week 14, Week 16, Week 20, Week 24 and Week 28
Efficacy and cutaneaous acceptability | Day 0, Week 4, Week 9, Week 12, Week 14, Week 16, Week 20, Week 24 and Week 28
  Questionnaire with 5 proposition for each question: completely agree, somewhat agree, neitheir agree or disagree, somewhat disagree, completely disagree

CONTACTS AND LOCATIONS:
Overall Officials: Gitanjali PETKAR, Dr, Principal Investigator — CIDP
Locations (1):
- CIDP, Phoenix, Mauritius

IPD SHARING:
Plan to Share IPD: No